CLINICAL TRIAL: NCT06437626
Title: Prospective International Multicenter Randomized, Double-blind, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of Mexidol® in Sequential Treatment of Patients in the Acute and Early Recovery Periods of Ischemic Stroke
Brief Title: Efficacy and Safety of Mexidol® in Stroke Therapy
Acronym: MIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MexidolMIR2023; PHS-APIS-004-MEX-SOL-TAB (Other: Ministry of Health, Russian Federation)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Neuroprotective Agents; Antioxidants; Stroke Rehabilitation; Recovery of Function; Brain Ischemia; Acute Stroke; Acute Cerebrovascular Accident; Cerebral Stroke; Neuroprotection; Mexidol; Ethylmethylhydroxypyridine Succinate
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia | interventions — emoxypine succinate; ethylmethylhydroxypyridine succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mexidol® (Experimental): Participants received Mexidol® IV 500 mg 2 times a day for 10 days, then Mexidol® FORTE 250 orally 250 mg 1 tablet 3 times a day for 60 days
  Interventions: Drug: Mexidol (Ethylmethylhydroxypyridine Succinate)
- Placebo (Placebo Comparator): Participants received Placebo matching Mexidol® IV 500 mg 2 times a day for 10 days, then Mexidol® FORTE 250 orally 250 mg 1 tablet 3 times a day for 60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexidol (Ethylmethylhydroxypyridine Succinate) — 50 mg/ml IV solution, 250 mg tablets
  Arms: Mexidol®
Drug: Placebo — Placebo IV solution, Placebo tablets
  Arms: Placebo

SUMMARY:
The main purpose of the clinical trial is to evaluate the efficacy and safety of Mexidol® in sequential treatment for patients in the acute and early recovery periods of ischemic stroke compared to placebo. The effect of adding Mexidol® to standard therapy on the degree of impairment of vital functions was assessed including the degree of disability (according to the Modified Rankin Scale, mRS), the severity of neurological symptoms (according to the National Institutes of Health Stroke Scale, NIHSS) and the level of mobility of patients (according to the Rivermead Mobility Index).

DETAILED DESCRIPTION:
As the main purpose of the clinical study is to evaluate safety and efficacy of a neuroprotector (Mexidol®), it was crucial to develop strict protocol requirements that would help to avoid the challenges of estimation of neuroprotective effect for stroke therapy. The current treatment options for stroke are still limited and do not take into account rehabilitation period and patients' further quality of life.

As per protocol requirements, 313 participants were screened, 304 participants met all comprehensive eligibility criteria, 25 participants dropped out during the clinical trial period. The Modified Rankin Scale (mRS) was selected as the most representative primary outcome measuring tool due to the adequate representation of functional outcome. Additionally, the neuroprotective efficacy of Mexidol® was assessed for its ability to reduce stroke-related neurologic deficit, to improve mobility after stroke and to influence cognitive impairment and mood disorder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of first-ever hemispheric ischemic stroke (codes ICD-10: I63.0 - I63.9) with the time from onset of a stroke <48 hours.
* CT or MRI evidences of clinical diagnosis and no evidences of hemorrhagic stroke/hemorrhagic transformation of ischemic stroke.
* The written informed consent form (ICF) is signed and personally dated by the participant or by an impartial witness (by a person who is independent of the trial and cannot be unduly influenced by the people involved with the trial and who attends the informed consent process).
* The Modified Rankin Scale (mRS) score ≥3.
* The National Institutes of Health Stroke Scale (NIHSS) score from 9 to 15 points.
* Negative pregnancy test for women of childbearing age.
* Willingness to use reliable methods of contraception, and/or abstinence, for the duration of therapeutic product exposure.
* The ability to understand the purpose of research, risks associated with the research intervention, obligations and consequences of research participation and their right of withdrawing consent any time during the study.

Exclusion Criteria:

* BMI (Body Mass Index) > 35.
* Recurrent or hemorrhagic stroke confirmed by CT/MRI.
* Hemorrhagic transformation of ischemic stroke.
* Parkinson's disease/parkinsonism.
* Progressive Multiple Sclerosis.
* Intractable Epilepsy.
* Demyelinating diseases of central nervous system.
* Hereditary and degenerative diseases of the central nervous system.
* Infectious diseases of central nervous system in medical history.
* Traumatic brain injury with severe neurocognitive impairment in medical history.
* Congenital malformations of the nervous system or any neurological disorders that can affect participant's capability (including cognitive and motor skills) to follow protocol procedures.
* Thrombolysis or thrombectomy treatment prior the enrollment.
* Medical history of severe allergies.
* Evidence of hypersensitivity reactions or intolerance associated with ethylmethylhydroxypyridine.
* Evidence of lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Acute surgical pathology.
* Evidence of clinically significant first identified disorder or disease that can affect participant's ability to participate in the clinical trial.
* Evidence of clinically significant severe disease/condition that can affect participant's ability to participate in the clinical trial: respiratory diseases, cardiovascular diseases (CVDs) including SAP ≥ 200 mm Hg and DAP ≥ 100 mm Hg, liver disease with elevation of ALT/AST > 2 × ULN, kidney disease (еGFR<30ml/min/1.73 m2), endocrine disorders and diseases, gastrointestinal diseases, pulmonary embolism (PE), deep vein thrombosis (DVT), floating thrombus, convulsive syndrome, uncontrolled hyperthermia, uncontrolled hyperglycemia.
* Medical history of severe mental disorder.
* Dementia of the Alzheimer type (DAT).
* Medical history of cancers within 5 years prior to enrollment.
* Medical history of alcohol/drug addiction.
* Pregnancy or breastfeeding.
* Prescription or use of prohibited medications within 2 weeks prior to enrollment.
* Positive HIV, syphilis, hepatitis B and C test.
* Positive COVID-19 test.
* Participation in another trial within 3 months prior to enrollment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Almaty City Hospital № 7, Almaty, Kazakhstan
- Russia (15):
  - Kazan City Hospital № 7, Kazan'
  - Kemerovo City Clinical Hospital № 11, Kemerovo
  - Research Institute - Regional Clinical Hospital № 1, Krasnodar
  - Federal Center for Brain and Neurotechnology, Moscow
  - Russian National Research Medical University n.a. N. I. Pirogov, Moscow
  - Rostov State Medical University, Rostov-on-Don
  - Alexandrovskaya Hospital, Saint Petersburg
  - St. Petersburg Clinical Hospital № 26, Saint Petersburg
  - City Hospital № 40 of Kurortny District, Saint Petersburg
  - Samara Regional Clinical Hospital n.a. V. D. Seredavin, Samara
  - Central Clinical Medical and Sanitary Unit n.a. V. A. Egorov, Ulyanovsk
  - Voronezh Regional Clinical Hospital № 1, Voronezh
  - Vsevolozhsk Clinical Interdistrict Hospital, Vsevolozhsk
  - Yaroslavl Clinical Hospital № 2 (ICU), Yaroslavl
  - Yaroslavl Clinical Hospital № 2, Yaroslavl
- The first clinic of the Tashkent Medical Academy, Tashkent, Uzbekistan

REFERENCES:
- [Background] Shamalov NA, Fedin AI, Rakhimbaeva GS, Nurguzhaev ES, Khasanova DR, Solovyova EY, Melnikova EV, Yanishevsky SN, Mashin VV, Pizova NV, Poverennova IE, Chuprina SE, Agafina AS, Roshkovskaya LV. [Results of the international multicenter randomized, double-blind, placebo-controlled clinical trial for the evaluation of the efficacy and safety of the sequential therapy with ethylmethylhydroxypyridine succinate in patients in the acute and early recovery periods of ischemic stroke (MIR)]. Zh Nevrol Psikhiatr Im S S Korsakova. 2025;125(8. Vyp. 2):40-53. doi: 10.17116/jnevro202512508240. Russian. PMID 40898634
- [Derived] Koltsov IA, Shchukin IA, Fidler MS, Glukhareva AP, Chubykin VI. [Multimodal antioxidant therapy in ischemic stroke: from MIR trial to bedside]. Zh Nevrol Psikhiatr Im S S Korsakova. 2025;125(12. Vyp. 2):64-71. doi: 10.17116/jnevro202512512264. Russian. PMID 41456191
- See also: Related Info — https://doi.org/10.17116/jnevro202512508240

RESULTS

PARTICIPANT FLOW:
Groups:
- Mexidol®: Participants received Mexidol® IV 500 mg 2 times a day for 10 days, then Mexidol® FORTE 250 orally 250 mg 1 tablet 3 times a day for 60 days
  Mexidol: 50 mg/ml IV solution, 250 mg tablets
- Placebo: Participants received Mexidol Placebo matching Mexidol® IV 500 mg 2 times a day for 10 days, then Mexidol® FORTE 250 orally 250 mg 1 tablet 3 times a day for 60 days
  Placebo: Placebo IV solution, Placebo tablets
Period: Overall Study
Arm/Group | Mexidol® | Placebo
Started | 152 | 152
Completed | 141 | 138
Not Completed | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mexidol® | Placebo | Total
Number analyzed (Participants) | 152 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.45 (7.88) | 62.61 (7.49) | 62.53 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 104 | 100 | 204
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 16 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 139 | 136 | 275
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uzbekistan | 10 | 10 | 20
  Kazakhstan | 10 | 10 | 20
  Russia | 132 | 132 | 264
Modified Rankin Scale (mRS) [Mean (Standard Deviation); unit: units on a scale] — The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke. Possible scores range from 0 (no symptoms at all) to 5 (dead).
  units on a scale | 3.90 (0.50) | 3.94 (0.48) | 3.92 (0.49)
Percentage of Subjects Having Modified Rankin Scale (mRS) Scores >3 (Higher Degree of Disability) [Count of Participants; unit: Participants] | 152 | 152 | 304
Percentage of Subjects Having Modified Rankin Scale (mRS) Scores 0-1 (Normal or Lower Degree of Disa [Count of Participants; unit: Participants] | 0 | 0 | 0
National Institutes of Health Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: units on a scale] — The NIHSS is a systematic assessment tool for a quantitative measure of stroke-related neurologic deficit. It is a 15-item neurologic examination stroke scale used to evaluate the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (severe stroke), with the minimum score being a 0 (no stroke symptoms).
  units on a scale | 9 [9 to 11] | 10 [9 to 10] | 9.5 [9 to 10.5]
Rivermead Mobility Index (RMI) [Median (Inter-Quartile Range); unit: units on a scale] — The Rivermead Mobility Index (RMI) is a hierarchical mobility scale used in neurological rehabilitation. It includes 15 items related to bed mobility, transfers, standing, walking, stair use, and running. Each response is scored yes or no with 1 point for each yes answer. The scores are summed with a range from 0 (poor mobility) to 15 (excellent mobility).
  units on a scale | 3 [1 to 5] | 3 [2 to 5.5] | 3 [1.5 to 5.5]
Montreal Cognitive Assessment (MoCA test) [Median (Inter-Quartile Range); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a 30-point validated scale that covers multiple cognitive domains including spatiotemporal orientation, sustained attention, visuospatial function, executive function, verbal memory, language, naming, and abstract thinking.
  units on a scale | 22 [19 to 24] | 22 [19 to 25] | 22 [19 to 24.5]
Hospital Anxiety and Depression Scale, domain ANXIETY (HADS-A) [Median (Inter-Quartile Range); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a brief self-report measure that was specifically designed to screen for distinct dimensions of anxiety and depression in nonpsychiatric hospital departments; somatic symptoms were excluded [22 point scale for each domain (Anxiety or Depression): min value 0, max value 21, higher scores mean a worse outcome].
  units on a scale | 6 [3 to 8] | 5 [3 to 8] | 5 [3 to 8]
Hospital Anxiety and Depression Scale, domain DEPRESSION (HADS-D) [Median (Inter-Quartile Range); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a brief self-report measure that was specifically designed to screen for distinct dimensions of anxiety and depression in nonpsychiatric hospital departments; somatic symptoms were excluded [22 point scale for each domain (Anxiety or Depression): min value 0, max value 21, higher scores mean a worse outcome].
  units on a scale | 6 [4 to 8] | 5 [3 to 8] | 5 [3 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modified Rankin Scale (mRS) Scores at the End of the Course of Therapy
Description: The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke. Possible scores range from 0 (no symptoms at all) to 5 (dead) [6 point scale: min value 0, max value 5, higher scores mean a worse outcome]. Change = (Visit 4, Day 71(+2) - Visit 0, Day 0-1 Scores).
Time Frame: Baseline, Day 71
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 141 | 138
score on a scale | -2.45 [-2.70 to -2.23] | -2.01 [-2.25 to -1.87]

2. Secondary Outcome: Percentage of Subjects Having Modified Rankin Scale (mRS) Scores >3 (Higher Degree of Disability) at the End of the Course of Therapy
Description: The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke. Possible scores range from 0 (no symptoms at all) to 5 (dead) [6 point scale: min value 0, max value 5, higher scores mean a worse outcome].
Time Frame: Day 71
Measure: Count of Participants; unit: Participants
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 141 | 138
Participants | 22 | 39

3. Secondary Outcome: Percentage of Subjects Having Modified Rankin Scale (mRS) Scores 0-1 (Normal or Lower Degree of Disability) at the End of the Course of Therapy
Description: as for outcome 2
Time Frame: Day 71
Measure: Count of Participants; unit: Participants
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 141 | 138
Participants | 85 | 57

4. Secondary Outcome: Change From Baseline in the National Institutes of Health Stroke Scale (NIHSS) Score at the End of the Course of Therapy
Description: The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (severe stroke), with the minimum score being a 0 (no stroke symptoms) [43 point scale: min value 0, max value 42, higher scores mean a worse outcome]. Change = (Visit 4, Day 71(+2) - Visit 0, Day 0-1 Scores).
Time Frame: Baseline, Day 71
Population: The number of participants assessed with this scale is 276 as it does not include the assessment of fatal outcomes, unlike the modified Rankin scale.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 139 | 137
score on a scale | -7 [-9 to -6] | -7 [-8 to -5]

5. Secondary Outcome: Change From Baseline in the Rivermead Mobility Index (RMI) Score at the End of the Course of Therapy
Description: The Rivermead Mobility Index (RMI) is a hierarchical mobility scale used in neurological rehabilitation. It includes 15 items related to bed mobility, transfers, walking, stair use, and running. The test is comprised of 14 questions, and the patient is then asked to stand for 10 seconds without any aid. Each response is scored yes or no with 1 point for each yes answer. The scores are summed with a range from 0 (poor mobility) to 15 (excellent mobility) [16 point scale: min value 0, max value 15, higher scores mean a better outcome]. Change = (Visit 4, Day 71(+2) - Visit 1, Day 1 Scores).
Time Frame: Baseline, Day 71
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 139 | 137
score on a scale | 10 [7 to 12] | 9 [7 to 11]

6. Secondary Outcome: Change From Baseline in the Montreal Cognitive Assessment (MoCA) Score at the End of the Course of Therapy
Description: The Montreal Cognitive Assessment (MoCA) is a 30-point validated scale that covers multiple cognitive domains including spatiotemporal orientation, sustained attention, visuospatial function, executive function, verbal memory, language, naming, and abstract thinking [31 point scale: min value 0, max value 30, higher scores mean a better outcome]. Change = (Visit 4, Day 71(+2) - Visit 1, Day 1 Scores).
Time Frame: Baseline, Day 71
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 139 | 137
score on a scale | 4 [2 to 6] | 3 [1 to 6]

7. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale Score, Domain ANXIETY (HADS-A), at the End of the Course of Therapy
Description: The Hospital Anxiety and Depression Scale (HADS) is a brief self-report measure that was specifically designed to screen for distinct dimensions of anxiety and depression in nonpsychiatric hospital departments; somatic symptoms were excluded [22 point scale for each domain (Anxiety or Depression): min value 0, max value 21, higher scores mean a worse outcome]. Change = (Visit 4, Day 71(+2) - Visit 1, Day 1 Scores).
Time Frame: Baseline, Day 71
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 139 | 137
score on a scale | -2 [-5 to 0] | -1 [-4 to 0]

8. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale Score, Domain DEPRESSION (HADS-D), at the End of the Course of Therapy
Description: as for outcome 7
Time Frame: Baseline, Day 71
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mexidol® | Placebo
Number analyzed (Participants) | 139 | 137
score on a scale | -2 [-4 to 0] | -1 [-4 to 0]

ADVERSE EVENTS:
Time Frame: Throughout the study [From Day 1 up to Day 71]
Arm/Group | Mexidol® | Placebo
All-Cause Mortality (participants affected / at risk) | 2/152 | 1/152
Serious Adverse Events (participants affected / at risk) | 6/152 | 4/152
Other Adverse Events (participants affected / at risk) | 36/152 | 39/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexidol® (N=152) | Placebo (N=152)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mexidol® (N=152) | Placebo (N=152)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
COVID-19 (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Latent syphilis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Blood pressure increased (Investigations) | 3 | 5
Blood pressure decreased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 2
Muscular weakness (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT06437626/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT06437626/SAP_001.pdf